CLINICAL TRIAL: NCT03438422
Title: Evaluation of the Impact of 3 Pollen Extracts in the Control of Urinary Incontinence in Women. Double-blind, Randomized, Placebo-controlled Study
Brief Title: Effect of Pollen Extract on Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Santiago Palacios (Other)
Responsible Party: Sponsor-Investigator, Dr. Santiago Palacios, Principal Investigator, Instituto Palacios
Organization: Instituto Palacios (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PJK-W10
Record Dates: First submitted 2018-02-08; First posted 2018-02-19 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Propolis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP A (Experimental): 1 tablet a day of pollen A extract containing (140 mg aqueous extract and 8mg lipid purified pollen, aqueous extract pumpkin seed 300mg, 10mg Vitamin E)
  Interventions: Dietary Supplement: Pollen extract
- GROUP B (Active Comparator): 1 tablet a day of pollen B extract containing (140 mg aqueous extract and lipid 8 mg of purified pollen)
  Interventions: Dietary Supplement: Pollen extract
- GROUP C (Active Comparator): 1 tablet a day of pollen extract C containing (Pollen extract 160 mg, pumpkin seed extract, 300 mg and Vitamin E 10 mg)
  Interventions: Dietary Supplement: Pollen extract
- PLACEBO (Placebo Comparator): 1 tablet a day of placebo
  Interventions: Dietary Supplement: Pollen extract

INTERVENTIONS:
Dietary Supplement: Pollen extract — 1 tablet a day

SUMMARY:
Study with food supplement to assess the eficacy of pollen extract on Urinary Incontinence

ELIGIBILITY:
Inclusion Criteria:

* Moderate, severe or very severe urinary incontinence, according to the severity index Incontinence Severity Index (ISI) * of Sandvik
* Healthy patients from 18 to 75 years of age
* Normal cytology in the last year and normal urological culture at inclusión
* Negative result in urine culture and normal vaginal canal (no evidence of dysplasia and / or infection)
* External vaginal area (vestibule and introitus) free of wounds or bleeding

Exclusion Criteria:

* Surgery for urinary incontinence
* Acute or recurrent infections of the urinary tract or genital infections (herpes or candida) in the last 3 months
* Malignant neoplasm or history of neoplasia in the last 5 years
* Concomitant disease such as a cardiac disorder, uncontrolled type I or II diabetes, lupus porphyria, relevant neurological disorders, any disease that in the opinion of the doctor could interfere with the treatment or resolution of the disease
* Anticoagulant alteration or thromboembolic alteration or taking anticoagulant drugs one week before treatment or during treatment for possible drug interaction (to allow inclusion, temporary cessation of use at the discretion of the doctor)
* History of immunosuppression or immunodeficiency (including HIV infection or AIDS) or use of immunosuppressive medications
* Hormonal imbalance, related to the thyroid, hypophysis or androgen not controlled
* Having a significant alteration in the areas under treatment or inflammatory alterations including but not limited to lacerations, abrasions or ulcers prior to treatment (time of resolution at the discretion of the doctor) or during treatment
* Dysplastic nevus in the treatment área
* Prolapse grade II according to the classification of the "Pelvic Organ Prolapse Quantification (ICS-POP-Q) System"
* Kegel exercises or electrostimulation at least 30 days before the start of treatment are not allowed

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 160 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Effect of the pollen extract on Urinary Incontinence | Baseline, two and three months
  To evaluate the effect of different pollen extracts on the number of leaks and on the amount of urine in each escape

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided